CLINICAL TRIAL: NCT05843903
Title: Teen Mom Study Feasibility Trial: A Multicomponent Digital Health Intervention to Improve Cardiometabolic Health in Pregnant Black Adolescents
Brief Title: Teen Mom Study Feasibility Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Collaborators: Mississippi State Department of Health (Other Government); Health Resources and Services Administration (HRSA) (U.S. Federal Agency); National Institute of General Medical Sciences (NIGMS) (NIH); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2022-110; P50MD017338 (NIH); U54GM115428 (NIH)
Record Dates: First submitted 2023-04-24; First posted 2023-05-06 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Physical Activity; Sedentary Behavior; Gestational Weight Gain; Social Determinants of Health
Keywords: implementation science; pragmatic clinical trial; telemedicine; health disparity, minority and vulnerable populations; behavior and behavior mechanisms; adolescent pregnancy; black maternal health
MeSH Terms: conditions — Motor Activity; Sedentary Behavior; Gestational Weight Gain; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- #BabyLetsMove (Experimental): There are four digital components to the intervention including Fitbit activity tracker, interactive self-monitoring and tailored feedback text messages, tailored skills training text messages and materials, and peer health coaching.
  Interventions: Behavioral: #BabyLetsMove

INTERVENTIONS:
Behavioral: #BabyLetsMove — The #BabyLetsMove digital health intervention uses a multi-level, systems-change approach. At the systems-level, racially concordant young adult WIC moms will be trained as health coaches. At the person level, adolescent WIC clients will be given empirically supported behavior goals, self-monitoring text messages with automated feedback, tailored skills training materials, a FitBit device, and tailored peer coaching support. The #BabyLetsMove intervention design is based on formative Teen Mom Study findings to build social cognition, affect, and skills to modify 3 concrete, achievable, and easily monitored behavioral targets: (1) Limit television viewing time to less than 2 hours per day; (2) Walk at least 10,000 steps per day; and (3) Do 20 minutes or more of exercise per day.

SUMMARY:
The proposed multicomponent digital health intervention has the potential to significantly impact the trajectory of maternal health in a rural, pregnant, Black adolescent population with the highest risks for cardiometabolic diseases worldwide. The proposed implementation strategy leverages mobile technologies which are ubiquitous across the socioeconomic gradient and proposes to train young adult WIC moms to deliver peer health coaching in a telehealth setting to address social barriers and support behavior change in pregnant, Black adolescent WIC clients in the Mississippi Delta - a rural region where the population is more than two-thirds percent Black and the teen birth rate is the highest in the United States. This is a scalable and sustainable approach to enhance WIC services and improve WIC's impact on population health and cardiometabolic health disparities in Black women.

DETAILED DESCRIPTION:
Teen Mom 2 will assess the feasibility, acceptability, and early efficacy of a 20-week multilevel, multicomponent digital health intervention, Mama Let's Move, delivered through the University of Mississippi Medical Center's Telehealth Center for Excellence in partnership with the Special Supplemental Nutritional Program for Women, Infants, and Children (WIC) to increase physical activity (PA) and reduce sedentary behavior (SB) in pregnant, Black adolescent WIC clients in the Mississippi Delta. The Social Ecological Model and TElehealth in CHronic Disease Model provide an empirical framework for considering multiple determinants of health behavior and evaluating mechanisms of implementation and intervention impacts. At the person level, pregnant, Black adolescent (15- to 19-years) WIC clients (n=20) will be given three empirically supported behavior goals to (1) watch 2 hours or less of television per day, (2) take 10,000 steps or more per day, and (3) engage in 20 minutes or more of organized exercise like prenatal yoga or dance videos per day. The intervention is designed to build social cognition, affect, and skills using four intervention components including a Fitbit activity tracker, interactive self-monitoring text messages with tailored feedback, tailored skills training text messages and materials, and peer health coaching. At the systems-level, racially concordant young adult (20- to 25-years) WIC moms (n=8) will be hired and trained to deliver peer health coaching in a telehealth setting to first, address social needs and second, to provide support for achieving the three behavior goals. The specific aims are to: (1) assess the impact of Mama Let's Move on objectively measured light-to-moderate PA and SB from baseline (<20-weeks' gestation) to 26- and 36-weeks' gestation in pregnant, Black adolescents; (2) use remote patient monitoring to objectively measure and characterize patterns of weight gain from baseline to 26- and 36-weeks' gestation; and (3) evaluate the feasibility and acceptability of training young adult WIC moms to provide health coaching in a telehealth setting. This study will advance public health and scientific knowledge in preparation for a future cluster randomized clinical trial by: training WIC moms to provide health coaching to pregnant, Black adolescents in a telehealth setting; developing an attention-control arm; assessing changes in adolescents' PA and SB throughout pregnancy in response to a 20-week intervention; characterizing patterns of weight gain throughout pregnancy in Black adolescents; comparing adolescents across counties and WIC providers; and evaluating an implementation partnership between WIC and the Telehealth Center of Excellence.

ELIGIBILITY:
Inclusion criteria:

* 15- to 19-years
* Black or African American
* <20 weeks' gestation
* Enrolled in WIC
* Residing in 1 of 8 Mississippi Delta Counties
* English speaking
* Own or have personal use of a mobile smart phone
* Singleton pregnancy
* Plan to carry the fetus to term and keep the infant after birth
* No history of chronic medical conditions in the past year that could influence weight loss or gain

Exclusion Criteria:

* Restrictions on physical activity or exercise

Ages: 15 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Acceptability | Perceptions of acceptability at 36 weeks' gestation (post-intervention)
  Qualitative interviews will be conducted with teens (n=20) to explore their satisfaction with the intervention components.
Appropriateness | Perceptions of appropriateness at study month 30 (of 36 months).
  Qualitative interviews will be conducted with peer health coaches (n=2) about their experience delivering coaching, case management support, and satisfaction with their role as a coach. Interviews with WIC leaders (n=3) and local WIC providers (n=5) will explore opinions on delivering coaching in a telehealth setting to enhance WIC's capacity to serve rural communities.
Intensity coaching session number | Average number of coaching sessions completed at 20 weeks (post-intervention)
  The intervention intensity will be determined based on the number of coaching sessions.
Intensity coaching session length | Average length in minutes of coaching sessions at 20 weeks (post-intervention)
  The intervention intensity will be determined based on the length in minutes of coaching sessions.
Intensity text message response number | Average number of text message responses at 20 weeks (post-intervention)
  The intervention intensity will be determined based on the number of responses to interactive text messages.

SECONDARY OUTCOMES:
Moderate-to-vigorous physical activity (MVPA) | Change in MVPA from baseline (< 16 weeks' gestation) to 26 weeks' gestation.
  GT9X ActiGraph accelerometer. Accelerometers will be worn on participants' non-dominant wrist for 7-days, 24-hours per day to record raw acceleration data using a sampling rate of 100 Hz that will be converted into objective measures. Counts: moderate (1952 - 5724 counts per minute) and vigorous (>5724 counts per minute) PA. Wear-time compliance will include 20 hours per day, > 4 days per week including 1 weekend day.
Sedentary behavior (SB) | Change in SB from baseline (< 16 weeks' gestation) to 26 weeks' gestation.
  GT9X ActiGraph accelerometer. Accelerometers will be worn on participants' non-dominant wrist for 7-days, 24-hours per day to record raw acceleration data using a sampling rate of 100 Hz that will be converted into objective measures. Counts: SB (<100 counts per minute). Wear-time compliance will include 20 hours per day, > 4 days per week including 1 weekend day.
Moderate-to-vigorous physical activity (MVPA) | Change in MVPA from baseline (< 16 weeks' gestation) to 36 weeks' gestation.
  GT9X ActiGraph accelerometer. Accelerometers will be worn on participants' non-dominant wrist for 7-days, 24-hours per day to record raw acceleration data using a sampling rate of 100 Hz that will be converted into objective measures. Counts: moderate (1952 - 5724 counts per minute) and vigorous (>5724 counts per minute) PA. Wear-time compliance will include 20 hours per day, > 4 days per week including 1 weekend day.
Sedentary behavior (SB) | Change in SB from baseline (< 16 weeks' gestation) to 36 weeks' gestation.
  GT9X ActiGraph accelerometer. Accelerometers will be worn on participants' non-dominant wrist for 7-days, 24-hours per day to record raw acceleration data using a sampling rate of 100 Hz that will be converted into objective measures. Counts: SB (<100 counts per minute). Wear-time compliance will include 20 hours per day, > 4 days per week including 1 weekend day.

CONTACTS AND LOCATIONS:
Overall Officials: Abigail Gamble, PhD, MS, Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gamble A, Beech BM, Blackshear C, Herring SJ, Welsch MA, Moore JB. Changes in Physical Activity and Television Viewing From Pre-pregnancy Through Postpartum Among a Socioeconomically Disadvantaged Perinatal Adolescent Population. J Pediatr Adolesc Gynecol. 2021 Dec;34(6):832-838. doi: 10.1016/j.jpag.2021.06.009. Epub 2021 Jul 13. PMID 34271198
- [Background] Gamble A, Beech BM, Blackshear C, Cranston KL, Herring SJ, Moore JB, Welsch MA. Recruitment planning for clinical trials with a vulnerable perinatal adolescent population using the Clinical Trials Transformative Initiative framework and principles of partner and community engagement. Contemp Clin Trials. 2021 May;104:106363. doi: 10.1016/j.cct.2021.106363. Epub 2021 Mar 15. PMID 33737198
- [Background] Gamble A, Saulters MM, Cranston KL, Jones DW, Herring SJ, Beech BM. Recruitment, Retention, and Engagement Strategies for Exercise Interventions With Rural Antenatal Adolescents: Qualitative Interviews With WIC Providers. J Public Health Manag Pract. 2020 Sep/Oct;26(5):497-502. doi: 10.1097/PHH.0000000000001027. PMID 32732725